CLINICAL TRIAL: NCT00027963
Title: The Efficacy Of Gabapentin In The Management Of Chemotherapy-Induced Peripheral Neuropathy: A Phase III Randomized, Double-Blind, Placebo-Controlled, Crossover Trial
Brief Title: Gabapentin in Treating Peripheral Neuropathy in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N00C3; CDR0000069098 (Registry Identifier: PDQ (Physician Data Query)); NCCTG-CCC-0020; NCI-P01-0196
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Neurotoxicity; Pain
Keywords: neurotoxicity; pain
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gabapentin (Experimental): Patients receive titrating doses of oral gabapentin twice daily and then three times daily for 3 weeks. Patients then receive a fixed dose of oral gabapentin three times daily for 3 weeks. Patients cross-over to therapy as in arm II at week 8.
  Quality of life is assessed at baseline and then at the end of weeks 6, 8, and 14.
  Interventions: Drug: gabapentin
- placebo (Placebo Comparator): Patients receive titrating doses of oral placebo and then a fixed dose of oral placebo as in arm I. Patients cross-over to therapy as in arm I at week 8.
  Quality of life is assessed at baseline and then at the end of weeks 6, 8, and 14.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: gabapentin
  Arms: gabapentin
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Gabapentin may be effective in relieving pain and other symptoms of peripheral neuropathy. It is not yet known if gabapentin is effective in treating peripheral neuropathy in cancer patients undergoing chemotherapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of gabapentin in treating pain and other symptoms of peripheral neuropathy in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether gabapentin improves the pain and other symptoms in cancer patients with chemotherapy-induced peripheral neuropathy.
* Determine the effect of this drug on symptom distress, mood states, functional abilities, and overall quality of life in these patients.
* Determine the toxic effects of this drug in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to neurotoxic chemotherapy (active vs nonactive and discontinued vs completed) and neurotoxic chemotherapeutic agents (vinca alkaloids vs taxanes vs platinum-based compounds vs combination of two or more of the above agents). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive titrating doses of oral gabapentin twice daily and then three times daily for 3 weeks. Patients then receive a fixed dose of oral gabapentin three times daily for 3 weeks. Patients cross-over to therapy as in arm II at week 8.
* Arm II: Patients receive titrating doses of oral placebo and then a fixed dose of oral placebo as in arm I. Patients cross-over to therapy as in arm I at week 8.

Quality of life is assessed at baseline and then at the end of weeks 6, 8, and 14.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Has received or is currently receiving neurotoxic chemotherapy, including taxanes (e.g., paclitaxel or docetaxel), platinum-based compounds (e.g., carboplatin, cisplatin, or oxaliplatin), or vinca alkaloids (e.g., vincristine or vinblastine)
* Pain or symptoms of peripheral neuropathy of at least 1 month duration attributed to chemotherapy-induced peripheral neuropathy

  * Average daily pain rating of at least 4 out of 10 using the pain numerical rating scale (where 0 is no pain and 10 is the worst pain possible) OR
  * Evidence of peripheral neuropathy of at least grade 1 out of 3 by ECOG Common

    * Toxicity Criteria for sensory neuropathy
* No other identified causes of painful paresthesia existing prior to chemotherapy

  * No radiotherapy-induced or malignant plexopathy
  * No lumbar or cervical radiculopathy
  * No pre-existing peripheral neuropathy of another etiology, including:

    * B12 deficiency
    * AIDS
    * Monoclonal gammopathy
    * Diabetes
    * Heavy metal poisoning
    * Amyloidosis
    * Syphilis
    * Hyperthyroidism or hypothyroidism
    * Inherited neuropathy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Life expectancy:

* At least 6 months

Renal:

* Creatinine no greater than 1.5 times upper limit of normal

Other:

* No prior allergic reaction or intolerance to gabapentin
* No significant psychiatric illness (e.g., mania, psychosis, or schizophrenia) that would preclude study compliance
* No extreme difficulty swallowing pills
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Other:

* More than 30 days since prior investigational agent for pain control
* Concurrent selective serotonin reuptake inhibitors allowed
* Concurrent nonsteroidal anti-inflammatory drugs allowed
* No concurrent tricyclic antidepressant (e.g., amitriptyline, nortriptyline, or desipramine)*
* No concurrent monoamine oxidase inhibitor*
* No concurrent opioid analgesic*
* No other concurrent adjuvant analgesic (e.g., anticonvulsant, clonazepam, or mexiletine)*
* No concurrent topical analgesics (e.g., lidocaine gel or lidocaine patch)*
* No concurrent amifostine
* No concurrent investigational agent for pain control NOTE: * For pain or symptoms due to chemotherapy-induced peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in pain and symptoms | Up to 14 weeks

SECONDARY OUTCOMES:
Quality of life | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (23):
- United States (22):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Rao RD, Michalak JC, Sloan JA, Loprinzi CL, Soori GS, Nikcevich DA, Warner DO, Novotny P, Kutteh LA, Wong GY; North Central Cancer Treatment Group. Efficacy of gabapentin in the management of chemotherapy-induced peripheral neuropathy: a phase 3 randomized, double-blind, placebo-controlled, crossover trial (N00C3). Cancer. 2007 Nov 1;110(9):2110-8. doi: 10.1002/cncr.23008. PMID 17853395